CLINICAL TRIAL: NCT05400655
Title: Safety and Efficacy of L9LS, a Human Monoclonal Antibody Against Plasmodium Falciparum, in an Age De-Escalation, Dose-Escalation Trial and a Randomized, Placebo-Controlled, Double-Blind Trial of Children in Western Kenya
Brief Title: Anti-malaria MAb in Kenyan Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); Kenya Medical Research Institute (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SERU 4413
Record Dates: First submitted 2022-05-12; First posted 2022-06-01 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Plasmodium Falciparum Infection; Malaria
Keywords: monoclonal; antibody; Kenya; malaria; children
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (22):
- Age de-escalation and dose-escalation study: Arm 1a: Age 5-10 years, 5 mg/kg of L9LS (Experimental): Healthy children aged 5-10 years receive a single dose of 5 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 2.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 1b: Age 5-10 years, Placebo (Placebo Comparator): Healthy children aged 5-10 years receive a single dose of placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 2.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 2a: Age 5-59 months, 5 mg/kg of L9LS (Experimental): Healthy children aged 5-59 months receive a single dose of 5 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 2b: Age 5-59 months, Placebo (Placebo Comparator): Healthy children aged 5-59 months receive a single dose of placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 2c: Age 5-10 years, 10 mg/kg of L9LS (Experimental): Healthy children aged 5-10 years receive a single dose of 10 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 2d: Age 5-10 years, Placebo (Placebo Comparator): Healthy children aged 5-10 years receive a single dose placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 3.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 3a: Age 5-10 years, 20 mg/kg of L9LS (Experimental): Healthy children aged 5-10 years receive a single dose of 20 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 4.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 3b: Age 5-10 years, Placebo (Placebo Comparator): Healthy children aged 5-10 years receive a single dose of placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 4.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 3c: Age 5-59 months, 10 mg/kg of L9LS (Experimental): Healthy children aged 5-59 months receive a single dose of 10 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 4.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 3d: Age 5-59 months, Placebo (Placebo Comparator): Healthy children aged 5-59 months receive a single dose of placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 4.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 4a: Age 5-59 months, 20 mg/kg of L9LS (Experimental): Healthy children aged 5-59 months receive a single dose of 20 mg/kg of L9LS one-time via subcutaneous administration.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 4b: Age 5-59 months, Placebo (Placebo Comparator): Healthy children aged 5-59 months receive a single dose of placebo via subcutaneous administration.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 5a: Age 5-71 months, 30 mg/kg of L9LS (Experimental): Healthy children aged 5-71 months receive a single dose of 30 mg/kg L9LS via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 6.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 5b: Age 5-71 months, Placebo (Placebo Comparator): Healthy children aged 5-71 months receive a single dose of placebo via subcutaneous administration. Once subjects reach day 7 post-administration without safety concerns dosing begins for arm 6.
  Interventions: Other: Placebo
- Age de-escalation and dose-escalation study: Arm 6a: Age 5-71 months, 40 mg/kg of L9LS (Experimental): Healthy children aged 5-71 months receive a single dose of 40 mg/kg L9LS via subcutaneous administration.
  Interventions: Drug: L9LS
- Age de-escalation and dose-escalation study: Arm 6b: Age 5-71 months, Placebo (Placebo Comparator): Healthy children aged 5-71 months receive a single dose of placebo via subcutaneous administration.
  Interventions: Other: Placebo
- Efficacy Study: Arm 1a: Age 5-17 months, 10-20 mg/kg of L9LS/Placebo (Experimental): Healthy children aged 5-17 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a single dose of placebo via subcutaneous administration.
  Interventions: Drug: L9LS; Other: Placebo
- Efficacy Study: Arm 1b: Age 5-17 months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS (Experimental): Healthy children aged 5-17 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a second single dose of 10-20 mg/kg L9LS via subcutaneous administration.
  Interventions: Drug: L9LS
- Efficacy Study: Arm 1c: Age 5-17 months, Placebo/Placebo (Placebo Comparator): Healthy children aged 5-17 months receive a single dose of placebo via subcutaneous administration. Six months later, participants receive a second single dose of placebo via subcutaneous administration.
  Interventions: Other: Placebo
- Efficacy Study: Arm 2a: Age 18-59 months, 10-20 mg/kg of L9LS/Placebo (Experimental): Healthy children aged 18-59 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a single dose of placebo via subcutaneous administration.
  Interventions: Drug: L9LS; Other: Placebo
- Efficacy Study: Arm 2b: Age 18-59 months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS (Experimental): Healthy children aged 18-59 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a second single dose of 10-20 mg/kg L9LS via subcutaneous administration.
  Interventions: Drug: L9LS
- Efficacy Study: Arm 2c: Age 18-59 months, Placebo/Placebo (Placebo Comparator): Healthy children aged 18-59 months receive a single dose of placebo via subcutaneous administration. Six months later, participants receive a second single dose of placebo via subcutaneous administration.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L9LS — Administered subcutaneously.
  Arms: Age de-escalation and dose-escalation study: Arm 1a: Age 5-10 years, 5 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 2a: Age 5-59 months, 5 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 2c: Age 5-10 years, 10 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 3a: Age 5-10 years, 20 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 3c: Age 5-59 months, 10 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 4a: Age 5-59 months, 20 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 5a: Age 5-71 months, 30 mg/kg of L9LS; Age de-escalation and dose-escalation study: Arm 6a: Age 5-71 months, 40 mg/kg of L9LS; Efficacy Study: Arm 1a: Age 5-17 months, 10-20 mg/kg of L9LS/Placebo; Efficacy Study: Arm 1b: Age 5-17 months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS; Efficacy Study: Arm 2a: Age 18-59 months, 10-20 mg/kg of L9LS/Placebo; Efficacy Study: Arm 2b: Age 18-59 months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS
Other: Placebo — Normal saline administered subcutaneously.
  Arms: Age de-escalation and dose-escalation study: Arm 1b: Age 5-10 years, Placebo; Age de-escalation and dose-escalation study: Arm 2b: Age 5-59 months, Placebo; Age de-escalation and dose-escalation study: Arm 2d: Age 5-10 years, Placebo; Age de-escalation and dose-escalation study: Arm 3b: Age 5-10 years, Placebo; Age de-escalation and dose-escalation study: Arm 3d: Age 5-59 months, Placebo; Age de-escalation and dose-escalation study: Arm 4b: Age 5-59 months, Placebo; Age de-escalation and dose-escalation study: Arm 5b: Age 5-71 months, Placebo; Age de-escalation and dose-escalation study: Arm 6b: Age 5-71 months, Placebo; Efficacy Study: Arm 1a: Age 5-17 months, 10-20 mg/kg of L9LS/Placebo; Efficacy Study: Arm 1c: Age 5-17 months, Placebo/Placebo; Efficacy Study: Arm 2a: Age 18-59 months, 10-20 mg/kg of L9LS/Placebo; Efficacy Study: Arm 2c: Age 18-59 months, Placebo/Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of one-time subcutaneous (SC) administration of monoclonal antibody (MAb) L9LS in healthy Kenyan children aged 5 months to 10 years, as well as the protective efficacy of one or two doses of L9LS against naturally occurring Plasmodium falciparum (Pf) infection among Kenyan children aged 5 to 59 months at enrollment, in a setting of perennial high transmission.

DETAILED DESCRIPTION:
A two-part, phase 2 trial evaluating the safety and tolerability of one-time subcutaneous (SC) administration of monoclonal antibody (MAb) L9LS in healthy Kenyan children aged 5 months to 10 years, as well as the protective efficacy of one or two doses of L9LS against naturally occurring Plasmodium falciparum (Pf) infection among Kenyan children aged 5 to 59 months at enrollment, in a setting of perennial high transmission.

Part 1 includes part 1a and part 1b and is an age de-escalation and dose-escalation study. In part 1a, in a stepwise fashion, children aged 5-10 years will receive 5 mg/kg of L9LS or placebo and be followed for 3 months to assess tolerability and safety. If acceptable tolerability and safety profiles are met at 1-week post-injection, the 5 mg/kg dose of L9LS or placebo will be administered to children aged 5-59 months while enrolling another cohort of children aged 5-10 years at a dose of 10 mg/kg of L9LS or placebo. If after 1 week, the 10 mg/kg dose is found to be safe in children aged 5-10 years and the 5 mg/kg dose is found to be safe in children aged 5-59 months, a 20 mg/kg dose of L9LS or placebo will be administered to children aged 5-10 years and a 10 mg/kg dose of L9LS or placebo to children aged 5-59 months. Finally, if these doses are found safe after 1 week, a 20 mg/kg dose of L9LS or placebo will be administered to children aged 5-59 months. Should tolerability and safety of all doses be acceptable in children aged 5-59 months, part 2 of the trial will begin. Part 1b of the study was added later and will include two additional dose escalation cohorts of children aged 5 to 71 months and will test 30 mg/kg L9LS and 40 mg/kg L9LS. Dosing in part 1 of the study will be weight-based and all doses will be administered SC in a double-blinded fashion. 12 participants in each age-dose group will be enrolled in a 3:1 ratio of L9LS to placebo, and all participants will be followed for a total of 3 months.

Part 2 is the efficacy study. Children 5-59 months of age will be randomized to receive a 10-20 mg/kg dose of L9LS or placebo by SC administration. There will be two L9LS cohorts, one 5-17 months of age and another 18-59 months of age, which will constitute one L9LS arm. A placebo arm will be composed of children 5-59 months of age. They will be followed over 12 months with monthly blood smear microscopy and polymerase chain reaction (PCR) and twice-monthly symptomatology and careseeking behavior questionnaires. Dosing will be based on three weight bands; all doses will be administered SC with fixed doses of 75 mg L9LS, 150 mg L9LS, or 225 Mg L9LS, resulting in a range of 10-20 mg/kg in a double-blinded fashion. Blood will be drawn to assess antibody titers at baseline, and at three additional time points over 12 months to establish pharmacokinetics (PK). Participants in the L9LS arm will be randomized 1:1 at baseline to receive either a second L9LS injection or a placebo injection to evaluate the additional efficacy of a second dose administered 6 months after the first dose. (Those in the placebo arm will receive a second injection of placebo.) Participants will be followed for an additional 6 months after the second injection with monthly blood smear microscopy and PCR, and a blood draw at month 11 to assess L9LS PK.

ELIGIBILITY:
Inclusion Criteria

Healthy children aged 5 months to 10 years (Part 1) or 5-59 months (Part 2). Weight ≥5 kg and weight ≤30 kg (Part 1) or weight ≥5 kg and ≤22.5 kg (Part 2) or weight ≥5 kg and ≤20 kg (for 30 mg/kg group) or weight ≥5 kg and ≤15 kg (for 40 mg/kg group), to ensure a maximum volume of two 2-mL (Part 1b) Hemoglobin level ≥8 g/dL. Height and weight Z-scores >-2. Living within Alego-Usonga sub-county. Able to participate for the duration of the trial. Parent and/or guardian of participant able to provide informed consent.

Exclusion Criteria

Individuals meeting any of the following criteria will be excluded from study participation:

Taking long-term cotrimoxazole. Participation or planned participation in any other interventional trial with an investigational product prior to the last required protocol visit or receipt of an investigational product within the past 30 days. (Note: Past, current, or planned participation in observational studies is NOT exclusionary.) Received any doses of any malaria vaccine. Participation in part 1 of this study (for individuals being screened for enrollment into part 2) Age < 12 months at the time the RTS,S/AS01 vaccine is anticipated to become available in the whole of Siaya County Current significant medical condition (neurologic, cardiac, pulmonary, hepatic, endocrine, rheumatologic, autoimmune, renal, oncologic, or hematological) or evidence of any serious underlying medical condition identified by medical history, physical examination, or laboratory examination.

Known sickle cell disease. (Note: Known sickle cell trait is NOT exclusionary.) White blood cell, absolute neutrophil, or platelet count outside the local laboratory-defined limits of normal. Subjects may be included at the investigator's discretion for values that are not clinically significant (ie., do not require any repeat or follow-up).

Alanine transaminase (ALT) or creatinine (Cr) level above the local laboratory-defined upper limit of normal. (Subjects may be included at the investigator's discretion for values that are not clinically significant.) Infected with HIV. History of a severe allergic reaction or anaphylaxis. Severe asthma (defined as asthma that is unstable or required emergency care, urgent care, hospitalization, or intubation during the past 2 years, or that has required the use of oral or parenteral corticosteroids at any time during the past 2 years).

Pre-existing autoimmune or antibody-mediated diseases including but not limited to: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, or autoimmune thrombocytopenia.

Known immunodeficiency syndrome. Use of chronic (≥14 days) oral or IV corticosteroids (excluding topical or nasal) at immunosuppressive doses (i.e., prednisone >10 mg/day) or immunosuppressive drugs within 30 days of day 0.

Known asplenia or functional asplenia. Clinical signs of malnutrition. Receipt of immunoglobulins and/or blood products within the past 6 months. Any history of menses. Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and comply with the study protocol.

Parental/guardian study comprehension examination score of <80% correct or per investigator discretion.

Receipt of a live vaccine or a killed vaccine within the past 2 weeks prior to study agent administration.

Known allergies or contraindication to dihydroartemisinin-piperaquine.

Use or known need at the time of pre-enrolment (DP administration) of concomitant prohibited medication, including:

Antimicrobial agents of the following classes (systemic use only):

Macrolides (e.g. erythromycin, clarithromycin, azithromycin, roxithromycin) Fluoroquinolones (e.g., levofloxacin, moxifloxacin, sparfloxacin) Pentamidine Antiarrhythmic agents (e.g. amiodarone, sotalol) Antihistamines (e.g. promethazine) Antifungals (systemic): ketoconazole, fluconazole, itraconazole Antiretrovirals: Saquinavir Diuretics (e.g. hydrochlorothiazide, furosemide) Antipsychotics (neuroleptics): haloperidol, thioridazine Antidepressants: imipramine, citalopram, escitalopram Antiemetics: domperidone, chlorpromazine, ondansetron Increased risk of salivary gland hypofunction (dryness of the mouth, swelling under the tongue and/or below the ear, halitosis) History of any other illness or condition which, in the investigator's judgment, may substantially increase the risk associated with the subject's participation in the protocol or compromise the scientific objectives, or other condition(s) that, in the opinion of the investigator, would jeopardize the safety or rights of a subject participating in the trial, interfere with the evaluation of the study objectives, or render the subject unable to comply with the protocol.

Ages: 5 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 912 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2024-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Titus Kwambai, MD, PhD, Principal Investigator — Centers for Disease Control and Prevention; Laura Steinhardt, PhD, MPH, Principal Investigator — Centers for Disease Control and Prevention; Peter D Crompton, MD, MPH, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID), National Institutes of Health (NIH)
Locations (1):
- Kenya Medical Research Institute (KEMRI) Center for Global Health Research (CGHR), Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers indefinitely after the completion of the primary endpoint by contacting one of the principal investigators.
Time Frame: Data may be requested at the time of publication or thereafter
Access Criteria: * De-identified data with approved outside collaborators under appropriate agreements.
  * De-identified results or data in publication and/or public presentations.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 912 children were consented
  * 233 screen failure
  * 58 late screen failures
  * 92 withdrew consent
  * 58 non-compliant
  * 15 study group complete
  * 35 eligible but not enrolled
  * 4 excluded due to other reasons
Period: Part 1A: Period 1
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Has Day 7 Data | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A: Period 2
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Has Day 7 Data | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up | 0 | 0 | 9 | 2 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 9 | 2 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A: Period 3
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Has Day 7 Data | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1A: Period 4
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Has Day 7 Data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1B/Part 2 - Period 1
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 54 | 54 | 54 | 54 | 52 | 56
Has Day 7 Data (Part 1B Only) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up (Part 1B Only) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Second Dose of Intervention (Efficacy Study Only) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 51 | 51 | 49 | 52 | 47 | 52
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 2 | 0 | 0 | 48 | 49 | 46 | 49 | 44 | 51
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 5 | 8 | 5 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 0 | 7 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0
Not completed — Missed multiple clinic visits | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 3
Period: Part 1B - Period 2
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Has Day 7 Data | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed Three Month Study Follow up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 1b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2d: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3b: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3d: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4b: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 5b: Age 5-71 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6b: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9LS/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo | Total
Number analyzed (Participants) | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 54 | 54 | 54 | 54 | 52 | 56 | 420
Age, Customized [Count of Participants; unit: Participants]
  5-120 months | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 54 | 54 | 54 | 54 | 52 | 56 | 420
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 6 | 0 | 7 | 1 | 4 | 1 | 3 | 3 | 6 | 2 | 5 | 1 | 1 | 1 | 28 | 34 | 27 | 29 | 27 | 27 | 222
  Male | 3 | 0 | 3 | 3 | 2 | 2 | 5 | 2 | 6 | 0 | 3 | 1 | 4 | 2 | 8 | 2 | 26 | 20 | 27 | 25 | 25 | 29 | 198
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black / Non-Hispanic | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 54 | 54 | 54 | 54 | 52 | 56 | 420
Region of Enrollment [Number; unit: participants]
  Kenya | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 54 | 54 | 54 | 54 | 52 | 56 | 420

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Adverse Events (AEs)
Description: Number of participants with at least one solicited local adverse events occurring within seven days of administration of intervention. Local reactogenicity included injection site pain, tenderness, bruising, swelling, redness, induration, pruritus, and other (e.g. injection site reaction). Adverse events were captured by Investigator examination and history from participants.
Time Frame: Age De-escalation and Dose escalation: within 7 days of administration of intervention; Efficacy study: within 7 days after first intervention, and 7 days after second intervention (second intervention occurred 6 months post first intervention)
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Groups:
- Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo: Healthy children aged 5-10 years receive a single dose of placebo via subcutaneous administration.
- Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo: Healthy children aged 5-59 months receive a single dose of placebo via subcutaneous administration.
  Placebo: Normal saline administered subcutaneously.
- Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo: Healthy children aged 5-71 months receive a single dose of placebo via subcutaneous administration.
  Placebo: Normal saline administered subcutaneously.
- Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS: Healthy children aged 5-17 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a second single dose of 10-20 mg/kg L9LS via subcutaneous administration.
  L9LS: Administered subcutaneously.
- Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS: Healthy children aged 18-59 months receive a single dose of 10-20 mg/kg L9LS via subcutaneous administration. Six months later, participants receive a second single dose of 10-20 mg/kg L9LS via subcutaneous administration.
  L9LS: Administered subcutaneously.
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 6 | 54 | 54 | 54 | 54 | 52 | 56
Participants
  Injection site pain | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Injection site swelling | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 1 | 2 | 0 | 0 | 1 | 1
  Injection site reaction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Injection site induration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Injection site pruritus | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injection site bruising | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Injection site redness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Local Adverse Events (AEs) (by Grade)
Description: The severity of local AEs was graded using the Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Clinical Trials Grade 1: Pain = does not interfere with activity; Tenderness = mild discomfort to touch; Erythema/Redness = 2.5-5 cm; Induration/Swelling = 2.5-5 cm and does not interfere with activity.
  Grade 2: Pain = Repeated use of non-narcotic pain reliever > 24 hours or interferes with daily activity; Tenderness= Discomfort with movement; Erythema/Redness = 5.1-10 cm; Induration/Swelling = 5.1-10 cm and interferes with activity.
  Grade 3: Pain = Any use of narcotic pain reliever or prevents daily activity; Tenderness = Significant discomfort at rest; Erythema/Redness = > 10 cm; Induration/Swelling = > 10 cm or prevents daily activity.
  Grade 4: Pain = Emergency room (ER) visit or hospitalization; Tenderness = ER visit or hospitalization; Erythema/Redness = Necrosis or exfoliative dermatitis; induration/Swelling = Necrosis Grade
  5: Death
Time Frame: as for outcome 1
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 6 | 54 | 54 | 54 | 54 | 52 | 56
Participants
  Grade 1 | 0 | 2 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 4 | 0 | 0 | 1 | 1 | 1 | 4 | 0
  Grade 2 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Systemic Adverse Events (AEs)
Description: Number of participants with local adverse events occurring within seven days of administration of intervention. Systemic reactogenicity events included pyrexia (fever), malaise (feeling unusually tired or unwell), muscle aches, headache, chills, nausea, and joint pain. Adverse events were captured by Investigator examination and history from participants.
Time Frame: as for outcome 1
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 6 | 54 | 54 | 54 | 54 | 52 | 56
Participants
  Chills | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Pyrexia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 4 | 12 | 13 | 7
  Malaise | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Muscle aches | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 6 | 4 | 3 | 6 | 5
  Joint pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Systemic Adverse Events (AEs) (by Grade)
Description: The severity of systemic adverse events occurring after the administration of L9LS was assessed using the grading scale below:
  Grade 1: Fever = 37.5^oC-37.9^oC; Fatigue, Headache, Myalgia = No interference with activity; Nausea = no interference with activity or 1-2 episodes/hour Grade 2: Fever = 38^oC-38.4^oC; Fatigue, Myalgia = Some interference with activity; Headache = Repeated use of non-narcotic pain reliever > 24 hours or some interference with activity; Nausea = Some interference with activity or > 2 episodes/24 hours Grade 3: Fever = 38.5^oC-39.5^oC; Fatigue = Prevents daily activity; Headache =Significant; any use of narcotic pain reliever or prevents daily activity; Myalgia =Significant; prevents daily activity; Nausea = Prevents daily activity, requires outpatient intravenous hydration Grade 4: Fever = > 39.5^oC; Fatigue, Headache, Myalgia = Emergency room (ER) visit or hospitalization; Nausea = ER visit or hospitalization for hypotensive shock
  Grade 5: Death
Time Frame: as for outcome 1
Population: Modified intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 6 | 54 | 54 | 54 | 54 | 52 | 56
Participants
  Grade 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 10 | 11 | 7 | 6 | 3 | 5
  Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 4 | 3 | 3 | 4 | 3
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Age De-escalation and Dose-escalation study: monitor for all adverse events (related & unrelated) till end of subject participation in study, which may be up to three months from dosing Efficacy study: Related adverse events - till end of subject participation in study, which may be up to 12 months from dosing Unrelated grade 1 or grade 2 adverse events - up to 28 days following dosing
Arm/Group | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 1/6 | 0/54 | 0/54 | 0/54 | 0/54 | 0/52 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/6 | 5/54 | 4/54 | 9/54 | 2/54 | 0/52 | 6/56
Other Adverse Events (participants affected / at risk) | 8/9 | 9/9 | 9/9 | 8/9 | 9/9 | 9/9 | 9/9 | 9/9 | 8/9 | 9/9 | 6/6 | 54/54 | 53/54 | 53/54 | 53/54 | 49/52 | 55/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo (N=9) | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo (N=9) | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo (N=6) | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo (N=54) | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS (N=54) | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo (N=54) | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo (N=54) | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS (N=52) | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo (N=56)
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Oesophageal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 2
Mumps (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Typhoid Fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Burns Second Degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
False Positive Investigation Result (Investigations) | 0 | 0 | 0 | 0 | NA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age De-escalation and Dose-escalation Study: Arm 1a: Age 5-10 Years, 5 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 2a: Age 5-59 Months, 5 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 2c: Age 5-10 Years, 10 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 3a: Age 5-10 Years, 20 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-10 Years, Placebo (N=9) | Age De-escalation and Dose-escalation Study: Arm 3c: Age 5-59 Months, 10 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 4a: Age 5-59 Months, 20 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-59 Months, Placebo (N=9) | Age De-escalation and Dose-escalation Study: Arm 5a: Age 5-71 Months, 30 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Arm 6a: Age 5-71 Months, 40 mg/kg of L9LS (N=9) | Age De-escalation and Dose-escalation Study: Age 5-71 Months, Placebo (N=6) | Efficacy Study: Arm 1a: Age 5-17 Months, 10-20 mg/kg of L9LS/Placebo (N=54) | Efficacy Study: Arm 1b: Age 5-17 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS (N=54) | Efficacy Study: Arm 1c: Age 5-17 Months, Placebo/Placebo (N=54) | Efficacy Study: Arm 2a: Age 18-59 Months, 10-20 mg/kg of L9LS/Placebo (N=54) | Efficacy Study: Arm 2b: Age 18-59 Months, 10-20 mg/kg of L9L/10-20 mg/kg of L9LS (N=52) | Efficacy Study: Arm 2c: Age 18-59 Months, Placebo/Placebo (N=56)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 8 | 8 | 4 | 4 | 1 | 3
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excessive Cerumen Production (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dental Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces Hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival Injury (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 4 | 8 | 5 | 5 | 6 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile Convulsion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling Hot (General disorders) | 2 | 1 | 3 | 1 | 1 | 5 | 2 | 2 | 2 | 1 | 0 | 6 | 3 | 6 | 10 | 8 | 6
Injection Site Induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection Site Swelling (General disorders) | 0 | 2 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 2 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 13 | 15 | 5 | 3 | 3 | 6
Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 2
Bacterial Infection (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 0
Body Tinea (General disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 4 | 2 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 5 | 0 | 3 | 3 | 2 | 1 | 2 | 8 | 2 | 4 | 3 | 5
Conjunctivitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysentery (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear Lobe Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Gastroenteritis (Infections and infestations) | 1 | 2 | 0 | 3 | 0 | 7 | 2 | 3 | 4 | 5 | 3 | 17 | 19 | 21 | 14 | 16 | 13
Gastroenteritis Salmonella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Helminthic Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 4 | 2 | 2 | 2 | 3 | 0 | 1 | 1 | 3 | 1 | 2 | 44 | 35 | 42 | 48 | 38 | 49
Mumps (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral Pustule (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 5 | 1 | 1
Otitis Media Acute (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 9 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 6 | 8 | 4 | 3 | 6 | 2
Rash Pustular (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 4 | 4 | 2 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5 | 4 | 6 | 4 | 5 | 2
Septic Rash (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 3 | 0
Tinea Capitis (Infections and infestations) | 1 | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 8 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 4 | 2 | 0 | 4 | 2 | 0 | 5 | 3 | 5 | 4 | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 9 | 8 | 7 | 4 | 9 | 8 | 8 | 7 | 7 | 5 | 36 | 33 | 34 | 36 | 38 | 36
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Viral Rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Wound Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accidental Exposure To Product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Greenstick Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 4 | 0 | 1 | 4
Headache (Nervous system disorders) | 0 | 1 | 2 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tonic Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Breast Enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital Pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus Genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 5 | 2 | 14 | 12 | 12 | 10 | 8 | 7
Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 3 | 1 | 0
Rash Vesicular (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT05400655/Prot_SAP_000.pdf